CLINICAL TRIAL: NCT05439876
Title: Getting SMART for Pediatric Epilepsy (Sleep, Melatonin, and Research Trial, SMART)
Brief Title: Getting SMART for Pediatric Epilepsy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202012143MIPC
Record Dates: First submitted 2022-06-20; First posted 2022-06-30 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Epilepsy in Children
MeSH Terms: interventions — Melatonin; Starch

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Melatonin (Experimental): Melatonin
  Interventions: Drug: Melatonin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — Melatonin 2 mg daily for 4 weeks
  Other Names: Melatonin supplement
  Arms: Melatonin
Drug: Placebo — Placebo daily for 4 weeks
  Other Names: Starch pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of melatonin for improving sleep in pediatric epilepsy.

DETAILED DESCRIPTION:
Sleep disturbances are more prevalent in children with epilepsy whose sleep can be disrupted by seizures occurring during the night and/or during the day. Melatonin is a naturally occurring hormone produced in the pineal which regulates sleep-wake cycles and facilitates quality sleep. Therefore, the purpose of this study is to evaluate the effect of melatonin for improving sleep in pediatric epilepsy.

ELIGIBILITY:
Inclusion Criteria:

- Children aged between 1 and 18 years with a confirmed diagnosis of epilepsy and with sleep problems

Exclusion Criteria:

* Children who are bedridden with limited mobility
* Children with liver or kidney dysfunction
* Children on hypnotics, antidepressants, or anxiolytics within 4 weeks before the baseline clinic visit
* Adolescent girls who are pregnant or breastfeeding
* Adolescent girls who have sexual activities but cannot take effective contraceptive measures during the trial

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 147 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Tso Lee, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Melatonin, Then Placebo: Participants first received melatonin (2 mg for children younger than 6 years or 4 mg for those 6 years and older) every night for 4 weeks. After a washout period of 2 weeks, they then received Placebo tablet each evening for 4 weeks.
- Placebo, Then Melatonin: Participants first received Placebo tablet every night for 4 weeks. After a washout period of 2 weeks, they then received Melatonin (2 mg for children younger than 6 years or 4 mg for those 6 years and older) every night for 4 weeks.
Period: First Intervention (for 4 Weeks)
Arm/Group | Melatonin, Then Placebo | Placebo, Then Melatonin
Started | 73 | 74
Completed | 64 | 64
Not Completed | 9 | 10
Period: Wash-out Period (for 2 Weeks)
Arm/Group | Melatonin, Then Placebo | Placebo, Then Melatonin
Started | 64 | 64
Completed | 64 | 64
Not Completed | 0 | 0
Period: Second Intervention (for 4 Weeks)
Arm/Group | Melatonin, Then Placebo | Placebo, Then Melatonin
Started | 64 | 64
Completed | 63 | 64
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Melatonin, Then Placebo: Melatonin First then Placebo
  Participants first received melatonin (2 mg for children younger than 6 years or 4 mg for those 6 years and older) every night for 4 weeks. After a washout period of 2 weeks, they then received Placebo tablet each evening for 4 weeks.
- Placebo, Then Melatonin: Placebo First then Melatonin
  Participants first received Placebo tablet every night for 4 weeks. After a washout period of 2 weeks, they then received Melatonin (2 mg for children younger than 6 years or 4 mg for those 6 years and older) every night for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Melatonin, Then Placebo | Placebo, Then Melatonin | Total
Number analyzed (Participants) | 73 | 74 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 73 | 74 | 147
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 34 | 68
  Male | 39 | 40 | 79
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Taiwan | 73 | 74 | 147
Sleep Onset Latency [Mean (Standard Deviation); unit: minutes] | 32.02 (22.06) | 29.65 (21.75) | 30.83 (21.84)

OUTCOME MEASURES:

1. Primary Outcome: Sleep Onset Latency
Description: Sleep onset latency was assessed by actigraphy.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 137 | 138
minutes | 22.80 (16.21) | 29.99 (29.74)

2. Secondary Outcome: Children's Sleep Disturbance
Description: Children's sleep disturbance was assessed by Children's Sleep Habits Questionnaire (CSHQ) total sleep disturbance score. There are 33 questions sumed as total score, range between 33 to 99. Higher score indicated more sleep disturbance problems in children.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Melatonin | Placebo
Number analyzed (Participants) | 137 | 138
score on a scale | 48.21 (6.71) | 49.41 (7.76)

ADVERSE EVENTS:
Time Frame: 14 weeks
Description: Six participants had a single non-serious adverse event each, evenly distributed between the melatonin (n=3) and placebo (n=3) groups. In the melatonin group, one participant reported mild hand weakness and decreased appetite. The other two participants in the melatonin group reported somnolence and fatigue. Adverse events in the placebo group included reported increased seizure frequency (n=1), body tremor (n=1), and agitation (n=1).
Arm/Group | Melatonin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/137 | 0/138
Serious Adverse Events (participants affected / at risk) | 0/137 | 0/138
Other Adverse Events (participants affected / at risk) | 3/137 | 3/138
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Melatonin (N=137) | Placebo (N=138)
mild hand weakness (Nervous system disorders) | 1 | 0
decreased appetite (Metabolism and nutrition disorders) | 1 | 0
somnolence and fatigue (Nervous system disorders) | 2 | 0
increased seizure frequency (Nervous system disorders) | 0 | 1
body tremors (Nervous system disorders) | 0 | 1
agitation (Nervous system disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT05439876/Prot_SAP_000.pdf